CLINICAL TRIAL: NCT02060461
Title: LASIK Flap Thickness and Visual Outcomes Using the WaveLight FS200 Femtosecond Laser: 3 Months Follow-up of Initial US Clinical Series
Brief Title: LASIK Flap Thickness and Visual Outcomes Using the WaveLight FS200 Femtosecond Laser
Acronym: FS200
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Cleveland Clinic (Other)
Collaborators: Alcon Research (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 11-744
Record Dates: First submitted 2013-12-16; First posted 2014-02-12 (Estimated); Results first posted 2018-03-23 (Actual); Last update posted 2018-03-23 (Actual); Status verified 2018-02

CONDITIONS: Myopia
MeSH Terms: conditions — Myopia

STUDY DESIGN:
Intervention Model Description: Contralateral eye study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- FS200 femtosecond laser LASIK (Experimental): LASIK flap created with an FS200 femtosecond laser system
  Interventions: Device: FS200 femtosecond laser LASIK
- IntraLase femtosecond laser LASIK (Experimental): LASIK flap created with an IntraLase femtosecond laser system
  Interventions: Device: IntraLase femtosecond laser LASIK

INTERVENTIONS:
Device: FS200 femtosecond laser LASIK
  Other Names: Alcon FS200 femtosecond laser
  Arms: FS200 femtosecond laser LASIK
Device: IntraLase femtosecond laser LASIK
  Other Names: AMO IntraLase femtosecond laser
  Arms: IntraLase femtosecond laser LASIK

SUMMARY:
The objective of this study is to evaluate the visual outcome, accuracy, predictability and complications of LASIK flap creation using the Alcon Wavelight FS200 Femtosecond laser and compare these results to those obtained using current IntraLase FS60 Femtosecond laser. The primary outcome to be evaluated is the flap thickness accuracy.

DETAILED DESCRIPTION:
Laser in situ keratomileusis (LASIK) is a method for treating myopia, hyperopia and astigmatism. In LASIK, the cornea is reshaped to focus images more clearly on the retina without the aid of glasses or contact lenses. LASIK involves two steps: creation of a corneal flap, which can be performed by a mechanical microkeratome or a femtosecond laser, and reshaping of the cornea by another laser, an excimer laser.

The accuracy of the LASIK flap thickness is a key safety consideration to reduce the likelihood of complications following LASIK. Femtosecond laser technology has significantly improved the predictability of LASIK flap dimensions while supporting similar visual acuity results.

The Alcon FS200 femtosecond laser is approved for human use by the United States Food and Drug Administration and was recently released in the US market. This study will directly compare outcomes of LASIK performed with this newer laser to those performed with the AMO IntraLase femtosecond laser.

ELIGIBILITY:
Inclusion Criteria:

* All patients with ametropia (Spherical, spherocylindrical, presbyopic) suitable for treatment by LASIK, including different target refractions (Plano or Monovision).

Exclusion Criteria:

* Patients unsuitable for LASIK procedure because of an estimated residual stromal bed < 300 microns after calculation of the ablation (Corneal thickness - flap thickness - simulated stromal ablation for the desired correction).
* Patients unsuitable for LASIK due suspicious topography for ectasia, form frust keratoconus or unstable ( more than 0.50 diopter change in sphere or cylinder in the last year) refraction.
* Patients with amblyopia or any eye disease that might limit the visual recovery.
* Patients younger than 18 years old.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2012-08; Primary Completion 2015-09 (Actual); Study Completion 2016-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: William J Dupps, MD, PhD, Principal Investigator — The Cleveland Clinic
Locations (1):
- Cleveland Clinic, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Rocha KM, Krueger RR. Spectral-domain optical coherence tomography epithelial and flap thickness mapping in femtosecond laser-assisted in situ keratomileusis. Am J Ophthalmol. 2014 Aug;158(2):293-301.e1. doi: 10.1016/j.ajo.2014.04.012. Epub 2014 Apr 30. PMID 24792107

RESULTS

PARTICIPANT FLOW:
Groups:
- Comparison of Femtosecond Lasers in LASIK: Outcomes of femtosecond-assisted LASIK will be compared between yes in subjects using the FS200 femtosecond laser in one eye and the IntraLase in the other.
Period: Overall Study
Arm/Group | Comparison of Femtosecond Lasers in LASIK
Started | 33
Completed | 33
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Comparison of Femtosecond Lasers in LASIK: Outcomes of femtosecond-assisted LASIK will be compared between yes in subjects using the FS200 laser in one eye and the IntraLase in the other.
Arm/Group | Comparison of Femtosecond Lasers in LASIK
Number analyzed (Participants) | 33
Age, Continuous [Mean (Standard Deviation); unit: years] | 30.5 (4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15
  Male | 18

OUTCOME MEASURES:

1. Primary Outcome: Evaluation of LASIK Flap Thickness
Description: Central LASIK flap thickness for each femtosecond laser. Each treatment was set for a 110 micrometer thick flap.
Time Frame: 3 months
Population: Contralateral eyes
Measure: Mean (Standard Deviation); unit: micrometers
Units Other Than Participants: eyes
Groups:
- FS200 Femtosecond Laser LASIK: FS200 laser used to create LASIK flap
- IntraLase Femtosecond Laser LASIK: IntraLase femtosecond laser used to create LASIK flap
Arm/Group | FS200 Femtosecond Laser LASIK | IntraLase Femtosecond Laser LASIK
Number analyzed (Participants) | 33 | 33
Number analyzed (eyes) | 33 | 33
micrometers | 105.8 (10.3) | 112.9 (8.2)
Statistical Analysis 1: Comparison: FS200 Femtosecond Laser LASIK vs IntraLase Femtosecond Laser LASIK; Paired Students t-test of FS200 and IntraLase intraoperative flap thickness measurements obtained by ultrasound pachymetry; Test type: Other; p = .003, t-test, 2 sided

ADVERSE EVENTS:
Groups:
- FS200 Femtosecond Laser LASIK: FS200 femtosecond laser used to create LASIK flap
- IntraLase Femotsecond Laser LASIK: IntraLase femtosecond laser used to create LASIK flap
Arm/Group | FS200 Femtosecond Laser LASIK | IntraLase Femotsecond Laser LASIK
All-Cause Mortality (participants affected / at risk) | 0/33 | 0/33
Serious Adverse Events (participants affected / at risk) | 0/33 | 0/33
Other Adverse Events (participants affected / at risk) | 0/33 | 0/33

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No